CLINICAL TRIAL: NCT02281409
Title: A Phase I/II Study of the Safety, Tolerability, and Immunoregulatory Activity of Mogamulizumab (KW-0761) in Subjects With Advanced and/or Metastatic Solid Tumors
Brief Title: Safety, Tolerability, and Immunoregulatory Activity of Mogamulizumab (KW-0761) in Subjects With Advanced and/or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 14-135
Record Dates: First submitted 2014-10-29; First posted 2014-11-03 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2020-12

CONDITIONS: Advanced Solid Tumors; Metastatic Solid Tumors
Keywords: Mogamulizumab (KW-0761); 14-135
MeSH Terms: interventions — mogamulizumab

ARMS (2):
- Phase I: Mogamulizumab (KW-0761) (Experimental): Patients will be enrolled to receive a weekly intravenous (IV) dose of KW-0761 ranging from 0.5 mg/kg to 10.0 mg/kg as feasible starting on Day 1 for 4 weeks. In the absence of toxicity or progression of disease, patients may continue receiving KW-0761 for up to 12 months. Subsequent treatment courses will consist of an infusion every other week. Following end of treatment or treatment completion date, a 24-week short term follow-up (STFU) period of observation will begin.
  Interventions: Biological: Mogamulizumab (KW-0761)
- Phase II: Mogamulizumab (KW-0761) (Experimental): Phase II of the study will enroll a total of 48 subjects, 16 patients in 3 tumor-specific expansion cohorts each treated at the RP2D (MTD, or highest dose tested in Phase I part of trial).
  Interventions: Biological: Mogamulizumab (KW-0761)

INTERVENTIONS:
Biological: Mogamulizumab (KW-0761)

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, KW-0761, an investigational drug, has on the patient and their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent form signed by the subject.
* Males and females 18 years or older at the time of dose initiation.
* Histologically confirmed unresectable solid tumor malignancy with at least 1 measurable lesion. In the expansion phase, eligibility will be limited to metastatic triple negative breast cancer that has received prior taxane and anthracycline therapy; Metastatic NSCLC that is not ALK+ and does not have a EGFR sensitizing mutation; and metastatic gastric cancer
* Previously treated for an advanced cancer and there are no curative therapy options available
* Karnofsky Performance Status ≥70 in the 30 day baseline period immediately prior to dosing.
* Evidence of adequate organ function by standard laboratory tests:

  * Serum creatinine (Cr) ≤1.5 X upper limit of normal (ULN)
  * Serum total and (T -Bil ) ≤1.5 X ULN (prior diagnosis or past history consistent with Gilbert's syndrome is an exception)
  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 X ULN
  * Platelets (Plts) ≥ 100,000/μl
  * Hemoglobin (Hgb) ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) ≥1000/mm3
* All female subjects of childbearing age must be either surgically sterile, postmenopausal for at least 1 year, or using an acceptable method of contraception. Examples of adequate methods of contraception include abstinence, intrauterine device, hormonal contraception, use of spermicide and a condom by sexual partner, or partner with a vasectomy. Adequate contraception must be used from the beginning of the screening period until at least 16 weeks after the last dose of KW-0761. Male subjects with partners of childbearing potential must use a barrier method of contraception from the day of the first dose of KW-0761 until at least 16 weeks after the last dose.
* Life expectancy > 12 weeks
* Previously treated for advanced cancer with no additional therapy options available known to prolong survival.

Exclusion Criteria:

* Evidence of clinically significant of central nervous system (CNS) metastases or symptomatic CNS metastases within 30 days prior to dosing.

History of autoimmune disease, except for vitiligo, diabetes, and autoimmune thyroiditis.

* A history of any major surgery within 6 weeks prior to dosing.
* Any history of systemic anticancer therapy (standard or experimental) completed within 30 days prior to dosing, with the exception of palliative ablation of lesion(s) as long as measurable disease lesion(s) remain for evaluation of exploratory endpoints.
* Any concomitant serious physical illness other than cancer (i.e., immune deficiency disease, bleeding disorder, etc.) within 1 year prior to dosing.
* Any history of Stevens-Johnson syndrome.
* Clinically significant heart disease, defined as NYHA Class III or IV.
* Any allergic reaction to a previously administered monoclonal antibody or other therapeutic protein.
* Any significant systemic infection within 4 weeks prior to dosing.
* Pregnancy or breast-feeding.
* An existing diagnosis of HIV, hepatitis B, hepatitis C, or any current laboratory findings or clinical signs and symptoms that suggest these conditions.
* Subjects with active herpes simplex or herpes zoster. Subjects with a history of herpes zoster who have had an outbreak within the last year will also be excluded. Subjects on prophylaxis for herpes who started taking medication at least 30 days prior to study entry, should continue to take the prescribed medication for the duration of the study.
* Unresolved immune- related adverse events following prior biological therapy
* Use of any investigational drugs within 30 days prior to dosing.
* Any condition that requires or is likely to require treatment with systemic corticosteroids within the Core Study Period and short term follow-up.
* Subjects that have had a myocardial infarction within the last 6 months.
* Subjects on any immunomodulatory drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-10; Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jedd Wolchok, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (0.5 mg/kg KW-0761 IV); Cohort 2 (1.0 mg/kg KW-0761IV) Q2W; Cohort 3 (3.0mg/kg KW-0761IV); Cohort 4 (10.0mg/kg KW-0761IV): Patients will be enrolled to receive a weekly intravenous (IV) dose of KW-0761 ranging from 0.5 mg/kg to 10.0 mg/kg as feasible starting on Day 1 for 4 weeks. In the absence of toxicity or progression of disease, patients may continue receiving KW-0761 for up to 12 months. Subsequent treatment courses will consist of an infusion every other week. Following end of treatment or treatment completion date, a 24-week short term follow-up (STFU) period of observation will begin. Phase II of the study will enroll a total of 48 subjects, 16 patients in 3 tumor-specific expansion cohorts each treated at the RP2D (MTD, or highest dose tested in Phase I part of trial).
  Mogamulizumab (KW-0761)
Period: Overall Study
Arm/Group | Cohort 1 (0.5 mg/kg KW-0761 IV) | Cohort 2 (1.0 mg/kg KW-0761IV) Q2W | Cohort 3 (3.0mg/kg KW-0761IV) | Cohort 4 (10.0mg/kg KW-0761IV)
Started | 3 | 3 | 5 | 6
Completed | 3 | 3 | 5 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (0.5 mg/kg KW-0761 IV) | Cohort 2 (1.0 mg/kg KW-0761IV) Q2W | Cohort 3 (3.0mg/kg KW-0761IV) | Cohort 4 (10.0mg/kg KW-0761IV) | Total
Number analyzed (Participants) | 3 | 3 | 5 | 6 | 17
Age, Continuous [Mean (Full Range); unit: years] | 55.3 [50 to 61] | 58.3 [24 to 80] | 57 [21 to 71] | 58.7 [42 to 72] | 58.7 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 3 | 6
  Male | 3 | 1 | 4 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 5 | 5 | 16
  Not Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 3 | 3 | 4 | 4 | 14
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 5 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: A standard 3+3 design will be utilized to determine the MTD. Four dose levels of KW-0761 will be investigated (0.5mg/kg, 1mg/kg, 3mg/kg, 10mg/kg). Patients will be treated in cohorts of size three to six and the dosage will be escalated if the clinical toxicity is acceptable.
Time Frame: 1 year
Measure: Number; unit: mg/kg KW-0761IV
Groups:
- Mogamulizumab (KW-0761): Patients will be enrolled to receive a weekly intravenous (IV) dose of KW-0761 ranging from 0.5 mg/kg to 10.0 mg/kg as feasible starting on Day 1 for 4 weeks. In the absence of toxicity or progression of disease, patients may continue receiving KW-0761 for up to 12 months. Subsequent treatment courses will consist of an infusion every other week. Following end of treatment or treatment completion date, a 24-week short term follow-up (STFU) period of observation will begin. Phase II of the study will enroll a total of 48 subjects, 16 patients in 3 tumor-specific expansion cohorts each treated at the RP2D (MTD, or highest dose tested in Phase I part of trial).
  Mogamulizumab (KW-0761)
Arm/Group | Mogamulizumab (KW-0761)
Number analyzed (Participants) | 22
mg/kg KW-0761IV | 10.0

2. Secondary Outcome: Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (0.5 mg/kg KW-0761 IV) | Cohort 2 (1.0 mg/kg KW-0761IV) Q2W | Cohort 3 (3.0mg/kg KW-0761IV) | Cohort 4 (10.0mg/kg KW-0761IV)
Number analyzed (Participants) | 3 | 3 | 5 | 6
Participants
  Progressive disease | 1 | 0 | 4 | 4
  Stable disease | 2 | 2 | 1 | 1
  Not entered | 0 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cohort 1 (0.5 mg/kg KW-0761 IV) | Cohort 2 (1.0 mg/kg KW-0761IV) Q2W | Cohort 3 (3.0mg/kg KW-0761IV) | Cohort 4 (10.0mg/kg KW-0761IV)
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 5/5 | 6/6
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 2/5 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (0.5 mg/kg KW-0761 IV) (N=3) | Cohort 2 (1.0 mg/kg KW-0761IV) Q2W (N=3) | Cohort 3 (3.0mg/kg KW-0761IV) (N=5) | Cohort 4 (10.0mg/kg KW-0761IV) (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 2 | 0 | 0 | 0
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (0.5 mg/kg KW-0761 IV) (N=3) | Cohort 2 (1.0 mg/kg KW-0761IV) Q2W (N=3) | Cohort 3 (3.0mg/kg KW-0761IV) (N=5) | Cohort 4 (10.0mg/kg KW-0761IV) (N=6)
Anemia (Blood and lymphatic system disorders) | 3 | 2 | 4 | 3
Lymphocyte count decreased (Investigations) | 3 | 3 | 3 | 5
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 2
Platelet count decreased (Investigations) | 1 | 1 | 0 | 1
White blood cell decreased (Investigations) | 1 | 2 | 0 | 3
Alkaline phosphatase increased (Investigations) | 1 | 0 | 3 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 3 | 2
Fatigue (General disorders) | 3 | 1 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1 | 4 | 4
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1
Skin & subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 1 | 0
Fibrinogen decreased (Investigations) | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1 | 2 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
INR increased (Investigations) | 1 | 0 | 1 | 2
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 2 | 0 | 0 | 0
Nail infection (Infections and infestations) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 2 | 1 | 1
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Serum amylase increased (Investigations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT02281409/Prot_SAP_000.pdf